CLINICAL TRIAL: NCT04754893
Title: Postbariatric EArly Discharge Controlled by Healthdot (PEACH)
Brief Title: Postbariatric EArly Discharge Controlled by Healthdot
Acronym: PEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICBE-2-36455
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-01

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Healthdot directly after surgery and leave the hospital on the same day (evening) (group A)
  Interventions: Device: Healthdot application
- Group b (No Intervention): Standard of care by staying one night in the hospital before returning home (group B)

INTERVENTIONS:
Device: Healthdot application — Healthdot device is applied on subject's chest after surgery
  Arms: Group A

SUMMARY:
This clinical investigation is a single center patient preference trial in a tertiary hospital in the Netherlands, designed to compare the outcome of two different recovery paths after standard of care bariatric surgery. The difference between both recovery paths is that half of the patients will get the standard of care by staying one night in the hospital before returning home (group B), while the other half will receive a Healthdot directly after surgery and leave the hospital on the same day (evening) (group A). 200 patients will be recruited and can choose whether they want to be assigned to the the regular recovery path or receive a Healthdot and leave the hospital on the same day. If they have no preference they will be randomly assigned to one of the two groups. Patients in the outpatient recovery group will wear the Healthdot for 7 days at home and vital signs (heart rate and respiratory rate, together with context data on activity and posture) will be transmitted to the hospital to monitor recovery. The study is mainly designed to investigate if the clinical outcome in both groups is equal (non-inferiority) based on a combined outcome measures like 30 days readmission rate and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult (equal or above 18)
* Approval for primary bariatric surgery (gastric sleeve or bypass) by a multidisciplinary bariatric team
* Willing and able to sign informed consent form
* Able to understand instructions
* In possession of a telephone on which patient can be reached for the duration of participation (day 1-8)
* An adult person must be present at the same location as the patient during the first night following surgery who is able to mobilize help or seek medical care if necessary.

Exclusion Criteria:

* Patients of psychiatric wards, inmates of prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Any skin condition, for example prior rash, discoloration, scars or open wounds at the area (Left lower rib) where the Healthdot needs to be placed
* Known allergy for the tissue adhesive used in the Healthdot (white band-aid)
* Use of topical that is known to influence the skin at the test area (such as medical and non-medical creams or lotions)
* Patient with active implantables such as Implantable Cardioverter Defibrilator (ICD) and pacemaker
* Expected participation less than 8 days
* Left lower rib (place where Healthdot will be applied) is involved in the area of surgery, area of disinfection or area where bandages are needed.
* Patients with antibiotic resitant infections (e.g. MRSA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Mortality | Within 30 days after primary surgery
  Mortality will be determined from the patient medical record
Severe postoperative complications (Clavien-Dindo IIIb or higher) | Within 30 days after primary surgery
  Severe postoperative complications will be determined from the patient medical record
Readmission (at least one night in hospital) | Within 30 days after primary surgery
  Readmission will be determined from the patient medical record
Mild complications (Clavien-Dindo II and IIIa) | Within 30 days after primary surgery
  Mild complications will be determined from the patient medical record
Prolonged length of stay (3 days or more in hospital) | Within 30 days after primary surgery
  Prolonged length of stay will be determined from the patient medical record

CONTACTS AND LOCATIONS:
Overall Officials: Simon Nienhuijs, Principal Investigator — Catharina Hospital, Eindhoven, The Netherlands
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Ede ES, Scheerhoorn J, Schonck FMJF, van der Stam JA, Buise MP, Nienhuijs SW, Bouwman RA. Lessons Learned from Telemonitoring in an Outpatient Bariatric Surgery Pathway-Secondary Outcomes of a Patient Preference Clinical Trial. Obes Surg. 2023 Sep;33(9):2725-2733. doi: 10.1007/s11695-023-06637-9. Epub 2023 Jul 7. PMID 37415024
- [Derived] Scheerhoorn J, van Ede L, Luyer MDP, Buise MP, Bouwman RA, Nienhuijs SW. Postbariatric EArly discharge Controlled by Healthdot (PEACH) trial: study protocol for a preference-based randomized trial. Trials. 2022 Jan 21;23(1):67. doi: 10.1186/s13063-022-06001-9. PMID 35063007